CLINICAL TRIAL: NCT02427854
Title: Can Perineal Tears and Obstetric Anal Sphincter Injuries in Palestine be Prevented? A Study of Two Different Interventions
Brief Title: Palestinian Perineum and Birth Complication Study
Acronym: PPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Croydon University Hospital (Other); University of Oslo (Other); Birzeit University Palestine (Unknown); University of Birmingham (Other)
Responsible Party: Principal Investigator, Erik Fosse, Professor, Head of Department, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2014/1727
Record Dates: First submitted 2015-03-09; First posted 2015-04-28 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2017-02

CONDITIONS: Complication of Labor and Delivery
Keywords: Major delivery complications; Perineal injuries; episiotomy
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No training (No Intervention): Incidence of obstetric perineal injuries in the participating hospitals before implementation of the manual perineal protection method.
- Education by animated training video (Active Comparator): Incidence of obstetric perineal injuries in the participating hospitals, after the delivery unit staff has been educated and trained to a perineal support by an animated training video only.
  Interventions: Behavioral: Education by animated training video
- Interactive hands on bedside training (Active Comparator): Incidence of obstetric perineal injuries in the participating hospitals, after the delivery unit staff has been educated and trained to a perineal support by an animated training video and additionally by an interactive hands-on bedside training.
  Interventions: Procedure: Interactive hands-on bedside training

INTERVENTIONS:
Behavioral: Education by animated training video — Training performed by watching an animated educational video.
  Arms: Education by animated training video
Procedure: Interactive hands-on bedside training — Training performed as a traditional bedside training supported by a trainer in person.
  Arms: Interactive hands on bedside training

SUMMARY:
In this study the investigators want to assess complications associated to pregnancy and delivery, and interventions used during labor.

Pregnancy and delivery related complications are a major health problem globally. Events during labor such as excessive bleeding, uterine rupture, emergency cesarean delivery; other instrumental deliveries and anesthesia problems are situations that potentially may lead to severe outcomes for the mother and child.

Diabetes, anemia and hypertensive disorders may also complicate both the pregnancy and delivery.

Between 60-80% of women delivering their first baby need suturing due to perineal tears (tears located to the area between the vagina and anus). Superficial perineal tears rarely cause long-term problems, but often lead to pain and discomfort immediately after birth. Deeper or severe perineal tears, involving the anal sphincter, may influence the woman's quality of life. This is mainly due to long-lasting pain, discomfort and sexual dysfunction, and the fact that obstetric anal sphincter tear is the main cause of anal incontinence. Recent clinical intervention studies have shown that the incidence of severe obstetric perineal tears may be reduced by 50-70% by introducing a bimanual support technique of the perineum. In these studies all midwives and gynecologists were trained in the bimanual support technique. When it comes to training in new medical techniques in general, some studies have shown that use of animated instructions on mobile phones may be a good alternative to the more traditional "hands-on" or "bedside" teaching methods. In a global perspective, it is important to study the efficacy of mobile units for transferring of new knowledge, especially for use in resource constrained settings.

DETAILED DESCRIPTION:
The main aim is to study the incidence of major delivery complications and perineal injuries during vaginal delivery in Palestine. A manual support technique of perineum will be introduced.

1. To assess the incidence of perineal tears, episiotomies, obstetric anal sphincter injuries and major obstetric complications in Palestine in a multicenter study involving three hospitals on the West Bank and three hospitals in Gaza.
2. To assess the present treatment of obstetric anal sphincter tears in Palestine.
3. To study whether intervention with bed-side training of the hands-on "the Norwegian-Finnish" support technique reduce the incidence of obstetric anal sphincter tears.
4. To study whether training by animated instructions of the same hands-on support technique, using smart phones or tablet computers, reduce the incidence of obstetric anal sphincter injuries.
5. To compare results between the two different training methods.
6. To study midwives' and doctors' attitudes towards "hands-on" training compared to training by animated instructions. The main aim is to assess the incidence of perineal injuries during vaginal delivery in Palestine, and to introduce a manual support technique of perineum. Norwegian intervention studies have shown that the incidence of obstetric anal sphincter injuries (OASIS) can be reduced by 40-70% by improving hands-on delivering techniques. The reduction was achieved by educating all staff on the delivery unit, implementing a new hands-on delivering technique. Some previous research has shown that non-interactive training by animated instructions or videos in emergency obstetric care, might be equally effective as conventional interactive hands-on training. However, the effectiveness of training by animated instructions compared to conventional training programs remains to be assessed properly. By performing a multicentre intervention study, the investigators will explore the effect of interactive hands-on training on the incidence of perineal injuries. Likewise the investigators will study effect of non-interactive training by animated instructions. Three hospitals on the West Bank (WB) and three in Gaza have accepted to participate. The investigators will also assess whether attitudes towards training methods influence the results.

The steps of observation, training and interventions in this study:

1. Intervention 1 (1 month):

   Education in diagnosis and repair of perineal injuries and implementation of system to register data.
2. Observation 1 (6 months):

   Data-registration baseline.
3. Intervention 2, (6 months):

   First part:

   In all participating hospitals, the training in hands-on manual perineal protection will be communicated by animated instruction accessible on tablet computers and smart phones. The information and instructions how to perform the manual perineal protection is transferred for the users by instruction video showing the method as an animation with voice-over in Arabic and English. All 6 hospitals implement this intervention simultaneously.

   Second part, the stepped wedge approach:

   After one month the first hospitals starts with the traditional bedside hands-on training of the midwives and physicians. Norwegian midwives and obstetricians support this training. The traditional bedside training then starts stepwise in the 6 hospitals, one month after each other, in a stepped wedge model.
4. Observation 2 (12 months):

There will be a one year observational period where all data is collected.

ELIGIBILITY:
Inclusion Criteria:

* all midwives and physicians working on labor ward in the participating hospitals.
* all women giving birth in the participating hospitals.
* both genders are included in the staff, and among the newborns

Exclusion Criteria:

* no exclusion criteria, the study aim is the education of the staff, and hospitals are compared as units.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51041 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of obstetric perineal injuries | 24 months
  All degrees of perineal injuries, including episiotomies, before and after intervention (education of the labour room staff)

SECONDARY OUTCOMES:
Occurrence of major delivery complications | 24 months
  Severe maternal complications during labor and delivery, such as excessive bleeding, uterine rupture, infections, seizures.
Occurrence of perineal injuries after education of the staff on diagnostics and repair | 24 months
  Effect of education on the anatomy of female pelvic floor, and a course on repair of injuries.

OTHER OUTCOMES:
Number of Participants with Adverse fetal outcome as a Measure of Safety and Tolerability | 24 months
  Adverse fetal outcome Morbidity and mortality of the fetus/newborn. Number of fetuses.
Number of participants with chronic diseases among delivering women in Palestine | 24 months
  Maternal pre-labor co-morbidity before pregnancy, during pregnancy and during delivery, such as diabetes, epilepsy, anemia, hypertensive conditions, medication.
Duration of delivery laboring women as a Measure of Safety and Tolerability | 24 months
  Duration of delivery
Number of Participants with obstetric intervention among laboring women in Palestine | 24 months
  Obstetric intervention during delivery
Number of Participants with operative deliveries among laboring women in Palestine | 24 months
  Operative delivery

CONTACTS AND LOCATIONS:
Overall Officials: Åse Vikanes, PhD, Study Director — Oslo University Hospital; Erik Fosse, PhD, Principal Investigator — Oslo University Hospital, University of Oslo
Locations (4):
- Palestinian Territories (4):
  - Palestinian Medical Complex, Ramallah, West Bank
  - AL Aqsa, Gaza
  - Shift, Gaza
  - Hebron, Hebron

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laine K, Pirhonen T, Rolland R, Pirhonen J. Decreasing the incidence of anal sphincter tears during delivery. Obstet Gynecol. 2008 May;111(5):1053-7. doi: 10.1097/AOG.0b013e31816c4402. PMID 18448735
- [Background] Laine K, Gissler M, Pirhonen J. Changing incidence of anal sphincter tears in four Nordic countries through the last decades. Eur J Obstet Gynecol Reprod Biol. 2009 Sep;146(1):71-5. doi: 10.1016/j.ejogrb.2009.04.033. Epub 2009 May 30. PMID 19482405
- [Background] Laine K, Skjeldestad FE, Sandvik L, Staff AC. Incidence of obstetric anal sphincter injuries after training to protect the perineum: cohort study. BMJ Open. 2012 Oct 17;2(5):e001649. doi: 10.1136/bmjopen-2012-001649. Print 2012. PMID 23075573
- [Background] Hals E, Oian P, Pirhonen T, Gissler M, Hjelle S, Nilsen EB, Severinsen AM, Solsletten C, Hartgill T, Pirhonen J. A multicenter interventional program to reduce the incidence of anal sphincter tears. Obstet Gynecol. 2010 Oct;116(4):901-908. doi: 10.1097/AOG.0b013e3181eda77a. PMID 20859154
- [Background] Raisanen S, Cartwright R, Gissler M, Kramer MR, Laine K, Jouhki MR, Heinonen S. Changing associations of episiotomy and anal sphincter injury across risk strata: results of a population-based register study in Finland 2004-2011. BMJ Open. 2013 Aug 17;3(8):e003216. doi: 10.1136/bmjopen-2013-003216. PMID 23955189
- [Background] Raisanen SH, Vehvilainen-Julkunen K, Gissler M, Heinonen S. Lateral episiotomy protects primiparous but not multiparous women from obstetric anal sphincter rupture. Acta Obstet Gynecol Scand. 2009;88(12):1365-72. doi: 10.3109/00016340903295626. PMID 19852569
- [Background] Laine K, Rotvold W, Staff AC. Are obstetric anal sphincter ruptures preventable?-- large and consistent rupture rate variations between the Nordic countries and between delivery units in Norway. Acta Obstet Gynecol Scand. 2013 Jan;92(1):94-100. doi: 10.1111/aogs.12024. Epub 2012 Dec 5. PMID 23034015
- [Background] Stedenfeldt M, Oian P, Gissler M, Blix E, Pirhonen J. Risk factors for obstetric anal sphincter injury after a successful multicentre interventional programme. BJOG. 2014 Jan;121(1):83-91. doi: 10.1111/1471-0528.12274. Epub 2013 May 20. PMID 23682573
- [Background] Raisanen S, Vehvilainen-Julkunen K, Gissler M, Heinonen S. Up to seven-fold inter-hospital differences in obstetric anal sphincter injury rates- A birth register-based study in Finland. BMC Res Notes. 2010 Dec 23;3:345. doi: 10.1186/1756-0500-3-345. PMID 21182773
- [Background] Raisanen S, Kancherla V, Kramer MR, Gissler M, Heinonen S. Placenta previa and the risk of delivering a small-for-gestational-age newborn. Obstet Gynecol. 2014 Aug;124(2 Pt 1):285-291. doi: 10.1097/AOG.0000000000000368. PMID 25004348
- [Background] Raisanen S, Kancherla V, Gissler M, Kramer MR, Heinonen S. Adverse perinatal outcomes associated with moderate or severe maternal anaemia based on parity in Finland during 2006-10. Paediatr Perinat Epidemiol. 2014 Sep;28(5):372-80. doi: 10.1111/ppe.12134. Epub 2014 Jun 17. PMID 24938307
- [Background] Al-Zirqi I, Stray-Pedersen B, Forsen L, Vangen S. Uterine rupture after previous caesarean section. BJOG. 2010 Jun;117(7):809-20. doi: 10.1111/j.1471-0528.2010.02533.x. Epub 2010 Mar 24. PMID 20236103
- [Background] Zimmo MW, Laine K, Hassan S, Bottcher B, Fosse E, Ali-Masri H, Zimmo K, Falk RS, Lieng M, Vikanes A. Exploring the impact of indication on variation in rates of intrapartum caesarean section in six Palestinian hospitals: a prospective cohort study. BMC Pregnancy Childbirth. 2022 Dec 2;22(1):892. doi: 10.1186/s12884-022-05196-8. PMID 36461037
- [Background] Hassan S, Laine K, Fosse E, Abu-Rmeileh NM, Ali-Masri HY, Zimmo M, Zimmo K, Vikanes A, Ismail KM. Induction Of Labor Among Singleton Pregnancies In Six Palestinian Governmental Hospitals: A Population-Based Cohort Study. Int J Womens Health. 2019 Nov 7;11:597-605. doi: 10.2147/IJWH.S215781. eCollection 2019. PMID 31807087
- [Background] Ali-Masri HY, Hassan SJ, Zimmo KM, Zimmo MW, Ismail KMK, Fosse E, Alsalman H, Vikanes A, Laine K. Evaluation of Accuracy of Episiotomy Incision in a Governmental Maternity Unit in Palestine: An Observational Study. Obstet Gynecol Int. 2018 Oct 29;2018:6345497. doi: 10.1155/2018/6345497. eCollection 2018. PMID 30510580
- [Background] Ali-Masri H, Hassan S, Fosse E, Zimmo KM, Zimmo M, Ismail KMK, Vikanes A, Laine K. Impact of electronic and blended learning programs for manual perineal support on incidence of obstetric anal sphincter injuries: a prospective interventional study. BMC Med Educ. 2018 Nov 12;18(1):258. doi: 10.1186/s12909-018-1363-3. PMID 30419884
- [Background] Zimmo MW, Laine K, Hassan S, Bottcher B, Fosse E, Ali-Masri H, Zimmo K, Sorum Falk R, Lieng M, Vikanes A. Caesarean section in Palestine using the Robson Ten Group Classification System: a population-based birth cohort study. BMJ Open. 2018 Oct 24;8(10):e022875. doi: 10.1136/bmjopen-2018-022875. PMID 30361403
- [Background] Zimmo K, Laine K, Fosse E, Zimmo M, Ali-Masri H, Zucknick M, Vikanes A, Hassan S. Episiotomy practice in six Palestinian hospitals: a population-based cohort study among singleton vaginal births. BMJ Open. 2018 Jul 16;8(7):e021629. doi: 10.1136/bmjopen-2018-021629. PMID 30012790
- [Background] Zimmo KM, Laine K, Fosse E, Zimmo M, Ali-Masri H, Bottcher B, Zucknick M, Vikanes A, Hassan S. Impact of animated instruction on tablets and hands-on training in applying bimanual perineal support on episiotomy rates: an intervention study. Int Urogynecol J. 2019 Aug;30(8):1343-1350. doi: 10.1007/s00192-018-3711-6. Epub 2018 Jul 14. PMID 30008080
- [Background] Ali-Masri H, Hassan S, Ismail K, Zimmo K, Zimmo M, Fosse E, Vikanes A, Laine K. Enhancing recognition of obstetric anal sphincter injuries in six maternity units in Palestine: an interventional quality improvement study. BMJ Open. 2018 Jun 19;8(6):e020983. doi: 10.1136/bmjopen-2017-020983. PMID 29921684
- [Background] Zimmo M, Laine K, Hassan S, Fosse E, Lieng M, Ali-Masri H, Zimmo K, Anti M, Bottcher B, Sorum Falk R, Vikanes A. Differences in rates and odds for emergency caesarean section in six Palestinian hospitals: a population-based birth cohort study. BMJ Open. 2018 Mar 2;8(3):e019509. doi: 10.1136/bmjopen-2017-019509. PMID 29500211
- [Background] Hassan S, Vikanes A, Laine K, Zimmo K, Zimmo M, Bjertness E, Fosse E. Building a research registry for studying birth complications and outcomes in six Palestinian governmental hospitals. BMC Pregnancy Childbirth. 2017 Apr 11;17(1):112. doi: 10.1186/s12884-017-1296-6. PMID 28399841
- [Background] Zimmo K, Laine K, Vikanes A, Fosse E, Zimmo M, Ali H, Thakar R, Sultan AH, Hassan S. Diagnosis and repair of perineal injuries: knowledge before and after expert training-a multicentre observational study among Palestinian physicians and midwives. BMJ Open. 2017 Apr 7;7(4):e014183. doi: 10.1136/bmjopen-2016-014183. PMID 28389490
- [Background] Ali HY, Vikanes A, Anti M, Hassan S, Ismail KM, Zimmo K, Zimmo M, Fosse E, Laine K. Evaluation of an animated instructional video as a training tool for manual perineum support during vaginal delivery. Int J Gynaecol Obstet. 2017 May;137(2):213-219. doi: 10.1002/ijgo.12115. Epub 2017 Feb 27. PMID 28171679